CLINICAL TRIAL: NCT03134521
Title: Population Pharmacokinetic Analysis of Daptomycin in Patients With Osteoarticular Infections
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0182
Record Dates: First submitted 2017-03-29; First posted 2017-05-01 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Bone Infection; Joint Infection
Keywords: bone and joint infection; daptomycin; population pharmacokinetics; Glycoprotein-P (PgP)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Daptomycin is validated as a treatment of bone and joint infections by the Infectious Disease Society of America. However, most of studies did not investigate daptomycin pharmacokinetics in this indication while it is known that efficacy and toxicity concentration studies show a close therapeutic margin.

Evaluation of P-Glycoprotein (P-gp), a transmembrane transport protein, has demonstrated its influence on the concentration and intracellular activity of daptomycin. Recent work has linked the genetic polymorphism of P-gp to the pharmacokinetics of daptomycin, which may explain inter-individual variability but requires further explorations. Previous studies demonstrated existence of interindividual variabilities as sex, renal function and p-glycoprotein polymorphism couple with an intraindividual variabilities unexplained yet.

A population approach will be used to determinate the pharmacokinetics factors, their intra and interindividual variabilities, the parameters associated to those variabilities (as the p glycoprotein).

The investigator's goal is to evaluate different posology and to try to increase daptomycin efficacy and security in bone and joint infection.

ELIGIBILITY:
Inclusion Criteria:

Patients

* having had a bone or joint infection, with or without implant,
* having an antibiotherapy with daptomycin between December 2012 and December 2016 at the Croix-Rousse hospital
* are at least 18 years old

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having bone or joint infection, with or without implant, having an antibiotherapy with daptomycin
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | Month 6

SECONDARY OUTCOMES:
Area under the concentration-time curve | up to 6 months
typical daptomycin clearance and volume of distribution in the population | Month 6
Mean daptomycine plasma clearance | Month 6
  (unit, liters per hour)
Mean daptomycine volume of distribution | Month 6
  (unit, liters)
Inter-individual coefficient of variation of daptomycin clearance | Month 6
  (unit, %)
Inter-individual coefficient of variation of daptomycin volume of distribution | Month 6
  (unit, %)
Intra-individual coefficient of variation of daptomycin clearance | Month 6
  (unit, %)
Intra-individual coefficient of variation of daptomycin volume of distribution | Month 6
  (unit, %)
influence of demographic and biological covariates on pharmacokinetics (e.g. : renal function, gender) | Month 6
  the influence of demographic and biological covariates on pharmacokinetics will be assessed statistically by using the Akaike Information Criterion (AIC, no unit). AIC = -2xLL + 2P, where LL is the log-likelihood computed by the population algorithm and P is the number of parameters in the model. A covariate will be considered as significant if it is associated with a decrease in the AIC value compared with the base model without covariate.
influence of p-glycoprotein pharmacogenetics on daptomycin pharmacokinetics | Month 6
  the influence of P-glycoprotein pharmacogenetics on pharmacokinetics will be assessed statistically by using the Akaike Information Criterion (AIC, no unit). AIC = -2xLL + 2P, where LL is the log-likelihood computed by the population algorithm and P is the number of parameters in the model. The P-glycoprotein genotype will be considered as significant if it is associated with a decrease in the AIC value compared with the base model without covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Principal Investigator — Hospices Civils de Lyon - Hopital de la Croix Rousse

REFERENCES:
- [Derived] Tuloup V, Millet A, Taricco A, Parant F, Ferry T, Goutelle S. Evaluation of Limited Sampling Strategies for Bayesian Estimation of Daptomycin Area Under the Concentration-Time Curve: A Short Communication. Ther Drug Monit. 2023 Aug 1;45(4):562-565. doi: 10.1097/FTD.0000000000001070. Epub 2023 Jan 2. PMID 36728573